CLINICAL TRIAL: NCT00654030
Title: Allogeneic Cellular Vaccine 1650-G for Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Allogeneic Cellular Vaccine 1650-G for Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edward Hirschowitz (Other)
Collaborators: Kentucky Lung Cancer Research Program (Other)
Responsible Party: Sponsor-Investigator, Edward Hirschowitz, Associate Professor of Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTN-0505; UKIRB 06-0716-F3R (Other: University of Kentucky); ULIRB 065.07 (Other: University of Louisville); CIRB 1079747 (Other: Commonwealth Cancer Center IRB)
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung Cancer Vaccine; Early Stage Lung Cancer; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1650-G Vaccine (Experimental): Patients receive 2 injections of 1650-G Vaccine given 4 weeks apart, for a total of 52 weeks on study.
  Interventions: Drug: 1650-G Vaccine

INTERVENTIONS:
Drug: 1650-G Vaccine — .6ml injection administered intradermally in the thigh at week 0 and week 4
  Other Names: 1650-G Allogeneic Cellular Vaccine

SUMMARY:
Rationale: Vaccines made from allogeneic tumor cells may help the body build an effective immune response to kill tumor cells.

The Purpose of this study is to evaluate the effects of a lung cancer vaccine in patients with Stage I or Stage II Non-Small Cell Lung Cancer (NSCLC) after completion of initial definitive therapies.

DETAILED DESCRIPTION:
The study is an open label investigation of the cellular vaccine called 1650-G. Patients receive 2 vaccine injections intradermally in the thigh given 4 weeks apart. Patients will be followed weekly after each vaccine injection and then monthly for 4 months. Patient follow-up continues with evaluations at 6 months and 1 year after receiving the first vaccine injection. Immunologic responses to the vaccine will be assessed from blood samples obtained at each visit following immunizations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage I or Stage II Non-Small Cell Lung Cancer
* Surgically resected at least 4 weeks ago but not more than 6 months ago
* Bronchoalveolar carcinomas allowed
* Completion of any chemotherapy or radiation given in conjunction with Surgery (neoadjuvant or adjuvant)
* No evidence of disease following initial therapy evidenced by a CXR, CT or PET scan within 6 weeks of enrollment
* ECOG performance status of 0 to 2
* Adequate organ and marrow function defined as follows:

  * Hemoglobin ≥9.0 gm/dL
  * Bilirubin < 2.5 x upper limit of normal
  * AST <2.5 x upper limit of normal
  * ALT <2.5 x upper limit of normal
  * Creatinine <3 mg/dL
* Women of childbearing potential must have a negative pregnancy test and be willing to use acceptable methods of contraception through week 16.

Exclusion Criteria:

* Cardiovascular disease defined as:

  * New York Heart Association Class III or IV (Section 19.2) congestive heart failure
  * hemodynamically significant valvular heart disease
  * myocardial infarction within the last six months
  * active angina pectoris
  * uncontrolled ventricular arrhythmias
  * stroke within one year
  * known cerebrovascular disease
* History of HIV, infectious hepatitis, or chronic immunosuppressive disease
* concurrent shorter courses of immunosuppressive medications during and for 16 weeks after study treatment
* History of an allergic reactions to any colony stimulating factor (GCSF, GMCSF)
* Female patients must not be pregnant or breastfeeding.
* History of participation in any investigational drug study within 4 weeks preceding initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Hirschowitz, MD, Study Chair — University of Kentucky; John R Yannelli, PhD, Study Chair — University of Kentucky; Goetz H Kloecker, MD, Principal Investigator — University of Louisville; Thomas R Baeker, MD, Principal Investigator — Commonwealth Cancer Center; Dattatraya S Prajapati, MD, Principal Investigator — Owensboro Medical Health System
Locations (4):
- United States (4):
  - Commonwealth Cancer Center, Danville, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Owensboro Medical Health System, Owensboro, Kentucky

REFERENCES:
- [Background] Hirschowitz EA, Foody T, Kryscio R, Dickson L, Sturgill J, Yannelli J. Autologous dendritic cell vaccines for non-small-cell lung cancer. J Clin Oncol. 2004 Jul 15;22(14):2808-15. doi: 10.1200/JCO.2004.01.074. PMID 15254048
- [Background] Hirschowitz EA, Hiestand DM, Yannelli JR. Vaccines for lung cancer. J Thorac Oncol. 2006 Jan;1(1):93-104. PMID 17409835
- [Result] Hirschowitz EA, Mullins A, Prajapati D, Baeker T, Kloecker G, Foody T, Damron K, Love C, Yannelli JR. Pilot study of 1650-G: a simplified cellular vaccine for lung cancer. J Thorac Oncol. 2011 Jan;6(1):169-73. doi: 10.1097/JTO.0b013e3181fb5c22. PMID 21150468

RESULTS

PARTICIPANT FLOW:
Groups:
- 1650-G Arm: Patients receive 2 injections of 1650-G Vaccine given 4 weeks apart
Period: Overall Study
Arm/Group | 1650-G Arm
Started | 12
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | 1650-G Arm
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Responding to the Vaccine
Description: The endpoint is immunologic response measured by IFN-ELISPOT. It will be reported as the percent of patients responding to vaccine (>2 Standard Deviation increase from baseline levels pre-vaccine). The number of individuals responding (> 2 SD change from baseline vaccine) will provide an approximation of biologic efficacy of the vaccine.
Time Frame: 16 weeks after vaccination
Measure: Count of Participants; unit: Participants
Groups:
- 1650-G ARM: 2 immunizations of 1650-G given 4 weeks apart
Arm/Group | 1650-G ARM
Number analyzed (Participants) | 11
Participants | 6

ADVERSE EVENTS:
Arm/Group | 1650-G Arm
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1650-G Arm (N=12)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1/1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthroplasty (Surgical and medical procedures) | 1/1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1650-G Arm (N=12)
Abdominal Cramps (Gastrointestinal disorders) | 1 (1)
Abnormal absolute nymphs (Blood and lymphatic system disorders) | 1 (1)
Abnormal Albumin (Blood and lymphatic system disorders) | 2 (3)
Abnormal Glucose (Blood and lymphatic system disorders) | 2 (4)
Abnormal hematocrit (Blood and lymphatic system disorders) | 1 (4)
Abnormal hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Abnormal percent lymphs (Blood and lymphatic system disorders) | 1 (1)
Abnormal platelets (Blood and lymphatic system disorders) | 1 (2)
Abnormal RBC (Blood and lymphatic system disorders) | 1 (3)
Abnormal WBC (Blood and lymphatic system disorders) | 1 (1)
Absent Pedal Pulses (Cardiac disorders) | 1 (1)
Achiness (General disorders) | 1 (1)
Achy Joints (Musculoskeletal and connective tissue disorders) | 1 (1)
Allergic Rhinitis (General disorders) | 1 (1)
Alopecia (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3)
B12 Deficiency (Blood and lymphatic system disorders) | 1 (1)
Bilirubin (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cyst removed left foot (Surgical and medical procedures) | 1 (1)
Decreased range of motion (left arm) (Musculoskeletal and connective tissue disorders) | 1 (1)
Statis Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Edema at Injection Site (Skin and subcutaneous tissue disorders) | 4 (4)
Elevated BUN (Blood and lymphatic system disorders) | 1 (1)
Elevated Creatinine (Blood and lymphatic system disorders) | 1 (1)
Elevated Glucose (Blood and lymphatic system disorders) | 1 (1)
Elevated Sodium (Blood and lymphatic system disorders) | 1 (1)
Enlarged Heart (Cardiac disorders) | 1 (1)
Episodic pain- left shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Faint wheeze - left lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Fever (General disorders) | 2 (2)
Flu-like Symptoms (General disorders) | 2 (2)
Headaches (Nervous system disorders) | 2 (2)
Hospitalization for Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot Flashes (Endocrine disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Hypopigmentation RT Thigh (Skin and subcutaneous tissue disorders) | 1 (1)
Induration - Left Thigh (Skin and subcutaneous tissue disorders) | 4 (4)
Induration- Right Thigh (Skin and subcutaneous tissue disorders) | 4 (4)
Injection Site Reaction- Left Thigh (Skin and subcutaneous tissue disorders) | 5 (5)
Injection Site Reaction- Right Thigh (Skin and subcutaneous tissue disorders) | 4 (4)
Insect Bite, Right Buttock (Skin and subcutaneous tissue disorders) | 1 (1)
Insomnia (General disorders) | 2 (3)
Intermittent incisional pain, right side of chest (General disorders) | 1 (1)
Itching at site of Insect bite (Skin and subcutaneous tissue disorders) | 1 (1)
Joint Aches (General disorders) | 1 (1)
Left Hip pain (General disorders) | 1 (1)
Left Shoulder Pain (General disorders) | 1 (1)
Leg Cramps (General disorders) | 1 (1)
Low/Abnormal Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Low/abnormal RBC (Blood and lymphatic system disorders) | 1 (1)
Mucosal Ulceration on Tongue (Skin and subcutaneous tissue disorders) | 1 (1)
Mucositis/Stomatitis, Pharynx (Gastrointestinal disorders) | 1 (1)
Muscle Weakness, whole body (General disorders) | 1 (1)
Musculoskeletal-other-strain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal Congestion/Stuffiness (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Necrosis, right buttock (Skin and subcutaneous tissue disorders) | 1 (1)
Neurological Complaint (Nervous system disorders) | 1 (1)
Pain at site of insect bite; right buttock (General disorders) | 1 (1)
Pain at Injection Site (General disorders) | 1 (1)
Pain-Gastrointestinal-abdomen (Gastrointestinal disorders) | 1 (1)
Pain in Right Breast (General disorders) | 1 (1)
Pain at Injection Site (Skin and subcutaneous tissue disorders) | 1 (1)
Pain in Left Arm (General disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post Nasal Drip (General disorders) | 1 (1)
Pretibial Edema (Musculoskeletal and connective tissue disorders) | 1 (2)
Pulmonary/Upper Respiratory System Infection (Infections and infestations) | 3 (5)
Redness at Injection site (Skin and subcutaneous tissue disorders) | 2 (2)
Restless Leg Syndrome (Nervous system disorders) | 1 (2)
Ringing in Ears (Ear and labyrinth disorders) | 1 (1)
Sebaceous keratosis right temple (Skin and subcutaneous tissue disorders) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Sinus Drainage (General disorders) | 1 (2)
Sinus Pressure (General disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Thigh Nodule/Erythema (Right Thigh) (Skin and subcutaneous tissue disorders) | 1 (1)
Thoracotomy Pain- left side (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrush (General disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study chair (Dr. Edward Hirschowitz) is only party available to disclose, discuss, or publish trial results or information concerning the trial after completion.